CLINICAL TRIAL: NCT03025451
Title: Retrospective Evaluation of Athens Complete Health Improvement Program (CHIP) Database
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, David Drozek, Assistant Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16X44
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight and Obesity
Keywords: nutrition; exercise; stress; gender; age; community support; cardiovascular disease; diabetes; hypertension; dyslipidemia; cholesterol; overweight; obesity; lifestyle
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Dyslipidemias; Overweight; Obesity; Motor Activity; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Complete Health Improvement Program (Experimental): Participants in The Complete Health Improvement Program
  Interventions: Behavioral: The Complete Health Improvement Program

INTERVENTIONS:
Behavioral: The Complete Health Improvement Program — CHIP focuses on food, diet, activity, exercise, stress management, by viewing videos, cooking demonstrations, discussion, and exercise. Intervention nurtures intelligent self-care through enhanced understanding of the epidemiology, etiology, and risk factors associated with chronic lifestyle related diseases. The primary focus is the consumption of plant-based whole foods, such as fresh fruits, vegetables, whole grains, legumes, and nuts. The goal was to keep dietary fat below 20% of total calories, daily intake of added sugar below 10 tsps, sodium below 2,000 mg, and cholesterol below 50 mg. High fiber food intake (>35 g/day) is encouraged, and flexibility exercises, a daily walk of 30 minutes or 10,000 steps and daily use of stress management techniques.
  Other Names: CHIP

SUMMARY:
Data from participants in Athens CHIP classes from May 2011 to present will be analyzed to evaluate the differences in outcomes based on: 1) gender, 2) age, 3) whether a household member participated in the class with them.

Participants had health screens before and after completing the class. The data from the health screens that will be utilized for comparison will include: body mass index (BMI), blood pressure, and fasting blood sugar and lipid levels.

DETAILED DESCRIPTION:
Identified data will be provided to the PI from Live Healthy Appalachia/CHIP on a flash drive. This data will be password protected by the research team. The data will consist of two different databases, 1) identifiers with health screen results, 2) identifiers with demographics (age, gender, household member in class). The researchers need data from both databases for this study. Each participant has been assigned a unique participant number by CHIP.

The databases will be combined by the research team, allowing the demographics to be matched to the biomarkers. The unique CHIP identifier will be maintained as a participant ID, while all other identifying data will then be deleted from the database.

The data will then be analyzed for relationships by a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in The Complete Health Improvement Program
* Signed the CHIP Request to Participate consent form, which includes the statement: "I understand that my test results are confidential but may be used for statistical analysis and group summaries."
* Completed both health screens

Exclusion Criteria: none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Weight | 4 months
  Weight

SECONDARY OUTCOMES:
Blood Pressure | 4 months
  Blood Pressure
Fasting Lipid Profile | 4 months
  Fasting Lipid Profile
Fasting Glucose | 4 months
  Fasting Glucose

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rankin P, Morton DP, Diehl H, Gobble J, Morey P, Chang E. Effectiveness of a volunteer-delivered lifestyle modification program for reducing cardiovascular disease risk factors. Am J Cardiol. 2012 Jan 1;109(1):82-6. doi: 10.1016/j.amjcard.2011.07.069. Epub 2011 Sep 23. PMID 21944675
- [Result] Leibold C, Shubrook JH, Nakazawa M, Drozek D. Effectiveness of the Complete Health Improvement Program in Reducing Risk Factors for Cardiovascular Disease in an Appalachian Population. J Am Osteopath Assoc. 2016 Feb;116(2):84-91. doi: 10.7556/jaoa.2016.020. PMID 26830523
- [Result] Vogelgesang J, Drozek D, Nakazawa M, Shubrook JH. Payer source influence on effectiveness of lifestyle medicine programs. Am J Manag Care. 2015 Sep 1;21(9):e503-8. PMID 26618437
- [Result] Drozek D, Diehl H, Nakazawa M, Kostohryz T, Morton D, Shubrook JH. Short-term effectiveness of a lifestyle intervention program for reducing selected chronic disease risk factors in individuals living in rural appalachia: a pilot cohort study. Adv Prev Med. 2014;2014:798184. doi: 10.1155/2014/798184. Epub 2014 Jan 16. PMID 24527219
- [Result] Kent LM, Morton DP, Rankin PM, Mitchell BG, Chang E, Diehl H. Gender differences in effectiveness of the Complete Health Improvement Program (CHIP) lifestyle intervention: an Australasian study. Health Promot J Austr. 2014 Dec;25(3):222-9. doi: 10.1071/HE14041. PMID 25476714